CLINICAL TRIAL: NCT02457858
Title: Manganese Porphyrin MnTE-2-PyP (BMX - 010) Preservation of Islet Cell Mass and Function for Clinical Islet Transplantation
Brief Title: Islet Isolation Using MnTE-2-PyP (BMX-010) - Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: BioMimetix Pharmaceutical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00045961
Record Dates: First submitted 2014-08-05; First posted 2015-05-29 (Estimated); Last update posted 2022-05-11 (Actual); Status verified 2016-09

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Islet Transplant
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — manganese tetrakis-(N-ethyl-2 pyridyl) porphyrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BMX-010 treated islets (Experimental): Islet isolation using BMX-010
  Interventions: Drug: Islet isolation using BMX-010

INTERVENTIONS:
Drug: Islet isolation using BMX-010 — BMX-010 will be used as a supplement in islet isolation process.
  Other Names: MnTE-2-PyP

SUMMARY:
In this study, the investigators hypothesize that the addition of antioxidant BMX-010 to perfusion solution, digestion solution and culture medium during islet isolation process, can lead to greater preservation of islet mass and metabolic function, such as improved islet yield, viability, and functional potency.

This pilot study will involve up to 10 participants from the islet transplant waiting list at the Clinical Islet Transplant Program. All participants will receive islets isolated with the medication BMX-010. This is to assess the primary safety of BMX-010 on pancreata and islets. BMX-010 will be used only in the islet isolation process, and will not be given to participants as medication.

DETAILED DESCRIPTION:
Islet Transplantation is a procedure used in people with difficult to control Type 1 Diabetes. Insulin producing cells (islets) are isolated from a deceased donor pancreas. After the cells are carefully isolated from the donor pancreas, the islets are transplanted into the recipient's liver. These transplanted islets may produce insulin.

One of the challenges with islet transplant is the death of some of the islet cells during isolation and storage while awaiting transplant. This is caused, in part, by inflammation and "oxidization" of the islet tissue. Oxidization is a process that causes chemical stress on living cells. We are looking for medications that would reduce inflammation, reduce oxidization and minimize cell death during the isolation process.

BMX-010 is a new drug that we believe will help fight oxidization. It is an antioxidant that has been shown in lab studies to help islet cells survive isolation and keep them healthy and functioning. BMX-010 has not been used in human islet transplants in Canada before this study. BMX-010 has been used once in a patient who needed his pancreas removed - the islets were isolated and treated with BMX-010, then transplanted back into the patient (auto-islet transplant). These results are promising and there have been no significant side-effects reported. There have also been studies using human islets, treated with BMX-010, transplanted into mice.

In this study, 10 patients will receive islets treated with BMX-010. This is to assess the primary safety of BMX-010 on pancreata and islets. For pancreata and islets treated with BMX-010, BMX-010 will be added in the steps of pancreas perfusion, pancreas digestion and islet culturing. Participants in the study will receive their islet transplants under standard of care islet transplant for all aspects of peri- and post-transplant management including immunosuppression. Islet transplant patients are followed as part of their standard of care, therefore the data collected for this study will be measured as part of routine clinical care, requiring no extra study specific clinic visits. We will review data collected up to day 30 post-transplant and will include the following: patient and graft survival data, biochemical data from routine blood work, routine and for cause imaging, metabolic testing, initiation of interventions to treat complications, and reporting of any adverse or serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

To be eligible the participant must have had type 1 diabetes mellitus (T1DM) for more than 5 years, complicated by at least 1 of the following situations that persist despite intensive insulin management efforts:

* a. Reduced awareness of hypoglycemia, as defined by the absence of adequate autonomic symptoms at plasma glucose levels < 3.0 mmol/L, indicated by, 1 or more episodes of severe hypoglycemia requiring third party assistance within 12 months, a Clarke score ≥4, HYPO score ≥1,000, lability index (LI) ≥400 or combined HYPO/LI >400/>300.
* b. Metabolic instability, characterized by erratic blood glucose levels that interfere with daily activities and or 1 or more hospital visits for diabetic ketoacidosis over the last 12 months.
* Participants must be capable of understanding the purpose and risks of the study and must sign a statement of informed consent.

Exclusion Criteria:

* 1. History of enrollment in any other islet transplant trials (at the discretion of the investigator).
* 2. Severe co-existing cardiac disease, characterized by any one of these conditions: (a) recent (within the past 6months) myocardial infarction; (b) left ventricular ejection fraction <30%; or (c) evidence of ischemia on functional cardiac exam.
* 3. Active alcohol or substance abuse, to include cigarette smoking (must be abstinent for 6 months prior to listing for transplant).
* 4. Psychiatric disorder making the subject not a suitable candidate for transplantation, (e.g., schizophrenia, bipolar disorder, or major depression that is unstable or uncontrolled on current medication).
* 5. History of non-adherence to prescribed regimens.
* 6. Active infection including Hepatitis C, Hepatitis B, HIV, or TB (subjects with a positive PPD performed within one year of enrollment, and no history of adequate chemoprophylaxis).
* 7. Any history of, or current malignancies except squamous or basal skin cancer.
* 8. BMI > 35 kg/m2 at screening visit.
* 9. Age less than 18 or greater than 68 years.
* 10. Measured glomerular filtration rate (GFR) <60 mL/min/1.73 m2.
* 11. Presence or history of macroalbuminuria (>300 mg/g creatinine).
* 12. Clinical suspicion of nephritic (hematuria, active urinary sediment) or rapidly progressing renal impairment (e.g. Increase in serum creatinine of 25% within the last 3-6 months).
* 13. Baseline Hb < 105g/L (<10.5 g/dL) in women, or < 120 g/L (<12 g/dL) in men.
* 14. Baseline screening liver function tests outside of normal range, with the exception of uncomplicated Gilbert's Syndrome. An initial LFT panel with any values >1.5 times the upper limit of normal (ULN) will exclude a patient without a re-test; a re-test for any values between ULN and 1.5 times ULN should be made, and if the values remain elevated above normal limits, the patient will be excluded.
* 15. Untreated proliferative retinopathy.
* 16. Positive pregnancy test, intent for future pregnancy or male subjects' intent to procreate, failure to follow effective contraceptive measures, or presently breast-feeding.
* 17. Evidence of significant sensitization on PRA (at the discretion of the investigator).
* 18. Insulin requirement >1.0 U/kg/day
* 19. HbA1C >12%.
* 20. Uncontrolled hyperlipidemia [fasting LDL cholesterol > 3.4 mmol/L (133 mg/dL), treated or untreated; and/or fasting triglycerides > 2.3 mmol/L (90 mg/dL)].
* 21. Under treatment for a medical condition requiring chronic use of steroids.
* 22. Use of coumadin or other anticoagulant therapy (except aspirin) or subject with PT/INR > 1.5.
* 23. Untreated Celiac disease.
* 24. Patients with Graves disease will be excluded unless previously adequately treated with radioiodine ablative therapy.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Islet yield using BMX-010, compared to current standard islet isolation data | Day -1 pre-transplant (Islet yield will be recorded as standard-of-care routine practice)
  To assess the safety of treating pancreata using BMX-010 prior to islet transplantation, treated islet isolation data will be measured and recorded, compared to current standard islet isolation data.

SECONDARY OUTCOMES:
Islet isolation quantity and quality using BMX-010, compared to current standard islet isolation data | Day -1 pre-transplant (Islet isolation quantity and quality will be recorded as standard-of-care routine practice)
  To demonstrate efficacy of BMX-010 to improve islet isolation quantity and quality prior to islet transplantation, treated islet isolation data will be measured and recorded, compared to current standard islet isolation data.
AE/SAE morbidity within 1 month post-transplant | up to 1 month post-transplant
  To demonstrate safety of BMX-010 in islet transplantation, Adverse Event/Serious Adverse Event morbidity within 1 month post-transplant will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: James Shapiro, MD PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- See also: Clinical Islet Transplant Program at University of Alberta — http://www.islet.ca